CLINICAL TRIAL: NCT00104949
Title: Phase II Study of Trastuzumab (NSC-688097) in Treatment of Locally Advanced or Metastatic Synovial Sarcoma
Brief Title: Trastuzumab in Treating Patients With Locally Advanced or Metastatic Synovial Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000413703; SWOG-S0346
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2006-12

CONDITIONS: Sarcoma
Keywords: adult synovial sarcoma; recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial | interventions — Trastuzumab

INTERVENTIONS:
Biological: trastuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Trastuzumab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well trastuzumab works in treating patients with locally advanced or metastatic synovial sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate (confirmed complete response and partial response) in patients with HER2/neu-overexpressing locally advanced or metastatic synovial sarcoma treated with trastuzumab (Herceptin^®).

Secondary

* Determine the frequency and severity of toxic effects of this drug in these patients.
* Determine overall survival and progression-free survival of patients treated with this drug.
* Correlate, preliminarily, SYT-SSX translocation, HER2/neu expression, and monophasic and biphasic phenotype with clinical outcomes in patients treated with this drug.

OUTLINE: This is a pilot, multicenter study.

Patients receive trastuzumab (Herceptin^®) IV over 90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 weeks until disease progression and then every 6 months for up to 2 years from study entry.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 10-40 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed synovial sarcoma meeting 1 of the following stage criteria:

  * Locally advanced disease, defined as 1 of the following:

    * Incurable by conventional multidisciplinary therapy, including surgery
    * Surgically resectable only with significant morbidity
  * Metastatic disease
* Tumor HER2/neu positive (2+ or 3+) by immunohistochemistry
* Tumor tissue must be available AND patient must be willing to allow specimen submission
* Measurable disease
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Hemoglobin > 8 g/dL
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)
* SGOT and/or SGPT < 1.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine < 1.5 times ULN OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* LVEF > 45% by MUGA

Gastrointestinal

* No active peptic ulcer disease
* No active gastrointestinal bleeding
* No active inflammatory bowel disease

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known HIV positivity
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent filgrastim (G-CSF)

Chemotherapy

* At least 3 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 60 days since prior radiotherapy to the target lesion*
* No concurrent radiotherapy NOTE: *Lesion must have demonstrated disease progression after completion of therapy

Surgery

* At least 21 days since prior major surgery and recovered

Other

* At least 60 days since prior embolization or radiofrequency ablation to the target lesion* NOTE: *Lesion must have demonstrated disease progression after completion of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Response rate (confirmed complete response and partial response)

SECONDARY OUTCOMES:
Progression-free survival at 1 and 2 years
Overall survival at 1 and 2 years
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ernest C. Borden, MD — The Cleveland Clinic; Rashmi Chugh, MD — University of Michigan Rogel Cancer Center; George D. Demetri, MD — Dana-Farber Cancer Institute; Margaret von Mehren, MD — Fox Chase Cancer Center; Vivien H.C. Bramwell, MB, BS, PhD, FRCP — Tom Baker Cancer Centre - Calgary; Karen H. Albritton, MD — Dana-Farber Cancer Institute